CLINICAL TRIAL: NCT07121335
Title: Cohort Study for Local Stereotactic Body Radiotherapy in Patients With Oligometastatic or Oligoprogressive Cancer
Brief Title: SMC Radiation Oncology SABR Cohort for Oligometastasis
Acronym: SABR-OMOP
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Nalee Kim, Assistant professor, Samsung Medical Center
Other Study IDs: SMC 2025-03-037
Record Dates: First submitted 2025-08-04; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Stereotactic Body Radiation Therapy (SBRT); Oligometastasis; Oligoprogression; ctDNA; Patient-Reported Outcomes (PRO)
Keywords: Stereotactic body radiotherapy; Oligometastasis; Oligoprogression; ctDNA
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Whole blood (20 mL) will be collected and retained for future DNA extraction and biomarker analyses, including circulating tumor DNA (ctDNA) profiling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — Stereotactic body radiotherapy (SABR) using photon or proton beams will be delivered per standard practice (1-5 fractions).

SUMMARY:
The goal of this observational study is to evaluate the efficacy and safety of stereotactic body radiotherapy (SABR) in patients with oligometastatic or oligoprogressive cancer.

The main questions it aims to answer are:

1. oncologic outcomes (progression-free survival, local failure rate),
2. patient-reported outcomes,
3. physician-assessed toxicity, and
4. dynamics of circulating tumor DNA (ctDNA) for biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Performance status (ECOG PS) 0-2
* Diagnosed with metastatic disease
* Confirmed to have oligometastatic/oligoprogressive cancer on imaging performed within 4 weeks (up to 5 lesions)

Exclusion Criteria:

* Patient with a history of prior radiotherapy to the site planned for SABR
* Patients with concomitant brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who are Confirmed to have oligometastatic/oligoprogressive cancer on imaging performed within 4 weeks (up to 5 lesions)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From start of SABR to the earliest of local failure, distant failure, death, or last follow-up. It will be measured at 1 month after completion of SABR, and at 6 months, 1 year, 2 years, and 3 years after SABR.
  Time from the start of stereotactic body radiotherapy (SABR) to the first documented event of local failure, distant failure, death from any cause, or last follow-up, whichever occurs first.
Physician assessed toxicity | 1 month after completion of SABR, and at 6 months, 1 year, 2 years, and 3 years after SABR.
  Evaluated by treating physician based on CTCAE ver 5.0
Patient-reported outcome | 1 month after completion of SABR, and at 6 months, 1 year, 2 years, and 3 years after SABR.
  It will be measured by PRO-CTCAE coreset 12.
Local failure | 1 month after completion of SABR, and at 6 months, 1 year, 2 years, and 3 years after SABR.
  Local regrowth or progression at the site of SABR.
Dynamics of ctDNA | It will be collected 1-week before SABR and 4-6 weeks after SABR.
  ctDNA analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No